CLINICAL TRIAL: NCT02292576
Title: Genetic and Epigenetic Mechanisms Underlying Cocoa Health Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11.21.NRC
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute dose/Chronic dose (Experimental): Acute dose/Chronic dose.
  Interventions: Other: Cocoa Pure; Other: Placebo
- Chronic dose/Acute dose (Experimental): Chronic dose/Acute dose.
  Interventions: Other: Cocoa Pure; Other: Placebo

INTERVENTIONS:
Other: Cocoa Pure — Cocoa Pure.
Other: Placebo — Placebo.

SUMMARY:
Evaluate if gene expression changes in SOD2 explain the health benefits of high polyphenols cocoa

DETAILED DESCRIPTION:
Evaluate if gene expression changes in SOD2 explain the health benefits of high polyphenols cocoa.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* BMI between 18.5 and 30 kg/m2
* Sedentary to moderate physical activity habits

Exclusion Criteria:

* Consumption of dietary supplements, antioxidants or anti-inflammatory medication, such as aspirin, ibuprofen, naproxen, or any medication that can affect the study outcomes
* Actively smoking
* Suspected abuse of alcohol or illicit drugs
* Significant illness within two weeks prior to study start or any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study
* Subject who cannot be expected to comply with study procedures
* Currently participating or having participated in another clinical trial during last 4 weeks prior to the beginning of this study
* Consumption of chocolate or its derivates 24 hours before the blood sample taken

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Measurement of changes in SOD2 gene expression | after acute dose and 4 weeks of chronic dose

SECONDARY OUTCOMES:
Determination of DNA methylation pattern in the chronic phase of the study | After 4 weeks of chronic dose
Evaluation of (-)epicatechin bioavailability in plasma | After 4 weeks of chronic dose
Determination of plasma antioxidant capacity as a marker of oxidative stress | After 4 weeks of chronic dose

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elizabeth Tejero Barrera, Ph.D., Principal Investigator — Instituto Nacional de Medicina Genomica